CLINICAL TRIAL: NCT01812694
Title: Lifestyle Interventions for Expectant Moms (LIFE-Moms) Phoenix
Brief Title: Lifestyle Interventions for Expectant Mothers (LIFE-Moms Phoenix) - Phoenix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999913055; 13-DK-N055
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-11

CONDITIONS: Obesity; Diet Therapy; Diabetes Type 2
Keywords: Pregnancy; Weight Control; Weight Gain
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard Care (Active Comparator): Standard prenatal care plus education
  Interventions: Behavioral: Enhanced standard care
- Intensive lifestyle intervention (Experimental): Intervention to limit excess gestational weight gain
  Interventions: Behavioral: Intensive lifestyle intervention

INTERVENTIONS:
Behavioral: Enhanced standard care — Standard prenatal care plus education
  Arms: Enhanced Standard Care
Behavioral: Intensive lifestyle intervention — Intervention to limit excess gestational weight gain
  Arms: Intensive lifestyle intervention

SUMMARY:
Background:

- LIFE-Moms (Lifestyle Interventions for Expectant Moms) is a national project that is studying pregnant women who are overweight or obese. It is looking at ways they can manage their weight gain in pregnancy and how this may affect them and their babies health at birth and through the first year. Researchers want to recruit pregnant women who are being treated at the Phoenix Indian Medical Center. They will participate in a two-part study.

Objectives:

- To study pregnant women who are in the LIFE-Moms project at the Phoenix Indian Medical Center.

Eligibility:

* Pregnant women at least 18 years of age who are overweight or obese.
* Participants must be receiving care at the Phoenix Indian Medical Center.
* Participants must be having only one child in their pregnancy (no twins or other multiple births).

Design:

* This study will have two parts. The first part will have three visits to obtain data about health early in pregnancy. It will also let participants and researchers find out if the participants are eligible and should continue in the second part of the study. In the second part, participants will be monitored throughout their pregnancy and during the first year after the baby s birth to test the effects of a lifestyle intervention to control weight gain during pregnancy.
* On the Part 1 study visits, participants will have a physical exam and medical history. They will provide blood, urine, hair, and other samples to be examined for possible genetic conditions.
* For the Part 2 study visits, participants will be placed in one of two treatment groups. Each group will receive the same prenatal and postnatal care that they would get if they did not join the study.
* The first group will have a lifestyle intervention program. They will spend about 2 hours every week with other members of their group to learn diet and activity behaviors that may help with their health.
* The second group will have an enhanced care program. They will be given additional information about health and pregnancy and be invited to attend three classes to learn about staying healthy during pregnancy.

DETAILED DESCRIPTION:
LIFE-Moms (Phoenix center) is a randomized clinical trial in overweight and obese pregnant women that will test the effects of an intensive lifestyle intervention on gestational weight gain, control of maternal hyperglycemia, and post-partum return to pre-pregnancy weight. The Phoenix center will be conducted in collaboration between the Phoenix Indian Medical Center (PIMC) nurse midwifery and obstetrics services and the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK). It is part of the LIFE-Moms Consortium consisting of six other clinical centers that will follow similar protocols and a research coordination unit.

American Indians are at high risk for developing obesity and type 2 diabetes mellitus (T2DM) and its complications. A major factor responsible for this finding is exposure of the fetus in the womb to its mother s diabetes, which increases the risk of diabetes in the offspring particularly during childhood and adolescence. This study is designed to evaluate the effects of an intensive lifestyle intervention (ILI) in at least 200 adult (age greater than or equal to 18 years) pregnant women who are eligible for prenatal care at PIMC. Interventions will be provided to overweight and obese pregnant women who do not have pregestational diabetes but may have (GDM), i.e., diabetes that first develops or is first recognized in pregnancy, or are at high risk of developing GDM. The lifestyle intervention will be patterned after the Diabetes Prevention Program (DPP) that prevented or delayed the onset of diabetes in non pregnant adults; the interventions will be modified to be appropriate in pregnancy. For women who develop diabetes, interventions will include coaching to optimize glycemic control.

Women will be randomly assigned to one of two intervention groups, assigned with equal probability: an enhanced standard of care group or an intensive lifestyle intervention group (ILI). Following delivery, all the mothers and infants will be treated in the same way regardless of their initial treatment group. For example, all mothers will be encouraged to breast feed and follow other recommended practices for the health of themselves and their babies. After delivery the mother will be invited to bring the infant to the research clinic five times during the first 6 months and again at 1 year of age. These follow up visits for the infant are timed 1) to understand the patterns of change in neonatal body composition and 2) to coincide, when possible, with well-child pediatric visits. We will also question the mothers and abstract data from the medical record regarding the child s feeding practice, overall health, hospitalizations, immunizations, and medicine use.

Outcomes will be assessed on the same schedule for both intervention groups. Prenatal measurements include demographic, anthropometric, and biochemical data. The latter will focus on periodic measures related to blood glucose (sugar), including glucose tolerance tests. Diet and physical activity will be assessed by questionnaires and objective activity monitors. Many of these tests will be repeated in the mother at 6-12 weeks and 12 months post-partum. Infant data at or shortly after birth and at months 1 through 6 and 12 will include weight, length, head size, estimated body fat, feeding practices, and medical record abstraction.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult pregnant women of any race or ethnicity may participate if they meet each of the following inclusion criteria:

1. At least 18 years of age.
2. Receive prenatal care at the nurse midwifery/obstetrics service of PIMC and plan to continue receiving such care throughout the pregnancy.
3. Able to have an OGTT prior to 16 weeks gestation. Hyperemesis can preclude some pregnant women from successfully completing the OGTT; these women will not be excluded if the fasting blood samples can be obtained.
4. Able to have an ultrasound examination to estimate fetal age.
5. Complete initial run-in screening visits to determine whether the woman can manage the tasks required of participation in an intensive intervention if randomized to the intervention group.
6. Able to commit the time required for the interventions and follow-up.
7. Singleton viable pregnancy. A twin pregnancy reduced to singleton before 14(0) weeks by project gestational age is acceptable. An ultrasound must be conducted before randomization that shows a fetal heartbeat; there should be no evidence of more than one fetus on the most recent pre-randomization ultrasound.
8. Gestational age at randomization no earlier than 9 weeks 0 days and no later than 15(6) weeks based on an algorithm that compares the LMP date and data from the earliest ultrasound.
9. Body mass index greater than or equal to 25 kilogram / square meter based on first trimester measured weight and on measured height. The earliest weight measurement before randomization, measured specifically for the study, will be used. Reported pre-pregnancy weight will not be used to determine eligibility because of the potential for inaccuracy. If the earliest weight measurement is conducted at 14(0) to 14(6) weeks or 15(0) to 15(6) weeks, 1 pound or 2 pounds will be subtracted from the measured weight, respectively, to adjust to a first trimester weight. This weight and the resultant BMI are defined as the baseline weight and BMI, respectively.

   EXCLUSION CRITERIA:
   * Diagnosis of diabetes prior to pregnancy or any of the following results of the oral glucose tolerance test at visit #1 that suggest diabetes prior to pregnancy: HbA1c greater than or equal 6.5 %, FPG greater than or equal 126 milligrams per deciliter, or 2-hour post-load plasma glucose greater than or equal 200 milligrams per deciliter (75 grams oral glucose tolerance test). All potential participants will have HbA1c and a 75 grams oral glucose tolerance test performed prior to randomization.
   * Women who meet the above criteria for diagnosed or presumed diabetes prior to pregnancy will be excluded. Others who meet criteria for GDM will be eligible. Criteria for GDM diagnosis will be based on ADA 2012 criteria (at least one of FPG greater than or equal to 92 milligrams per deciliter, 1 hour PG greater than or equal 180 milligrams per deciliter, or 2 hour PG greater than or equal to 153 milligrams per deciliter.)
   * Known fetal anomaly
   * Planned termination of pregnancy
   * History of three or more consecutive first trimester miscarriages
   * Past history of anorexia or bulimia by medical history or patient report. Binge eating disorder (BED) is not an exclusion.
   * Current eating disorder diagnosed by EDE-Q questions 2-4 and confirmed after discussion with the participant by study staff
   * Actively suicidal defined as a value greater than or equal 2 on the BDI-II question 9
   * Prior or planned (within 1 year of expected delivery) bariatric surgery
   * Current use of one or more of the following medications:

     * Metformin
     * Systemic steroids
     * Antipsychotic agents (e.g., Abilify (apriprazole), Haldol (haloperidol), Risperdal (resperidone), Seroquel (quetipapine), Zyprexa (olanzapine))
     * Anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight (e.g., Depakote (valproic acid), Lamictal (lamotrigine), Lithium, Neurontin (gabapentin), Tegretol (carbamazepine), Topamax (topiramate), Keppra (levetiracetam)
     * Medications for ADHD including amphetamines and methylphenidate
     * Any teratogenic agent Class D or X (site specific)
   * Continued use of weight loss medication including OTC and dietary supplements for weight loss (e.g., Adipex (phentermine), Suprenza(phentermine) Tenuate (dietheylpropion), Xenical (orlistat), Alli (orlistat), conjugated linoleic acid, Hoodia, Green tea extract, Guar gum, HydroxyCut, Sensa, Corti-slim, Chromium, chitosan, Bitter orange)
   * Contraindications to aerobic exercise in pregnancy specified in the ACOG Committee Opinion #267, 2002

     * Hemodynamically significant heart disease defined as an AHA class II (short of breath with exercise) or greater
     * Restrictive lung disease (e.g. pulmonary fibrosis)
     * Poorly controlled hyperthyroidism
     * Poorly controlled seizure disorder
     * Poorly controlled hypertension defined as a blood pressure greater than or equal 160/110 millimeters of mercury
     * History of extreme sedentary lifestyle (e.g. bed bound)
     * Orthopedic limitations to aerobic exercise
     * Severe anemia defined as a hemoglobin less than 8 grams per deciliter
     * Any condition that requires follow-up at specialty care clinics outside of PIMC (e.g., pregnancies at high risk for maternal or fetal demise)
   * Participation in another interventional study that influences weight control
   * Enrollment in this trial in a previous pregnancy
   * Intention of the participant or of the care provider for the delivery to be outside the greater Phoenix metropolitan area.
   * Participant s unwillingness or inability to commit to a 1 year follow-up of herself or her child, including planning to move away.
   * Inability or unwillingness to provide informed consent, in the English language, including consent for study staff to abstract data from all prenatal and delivery records (for the current pregnancy) whether the care or delivery occur at PIMC or elsewhere. English is the common language of the participants who receive care at PIMC. Some also speak tribal languages or Spanish. English is the language used in the intervention materials, the screening forms, and online documents. English is also the primary language of study staff.
   * Any condition that in the opinion of the investigators would interfere with consent, treatment or follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 36 weeks
  Weight at 36 weeks minus weight at baseline, kg

SECONDARY OUTCOMES:
Gestational Diabetes | 24-28 weeks gestation, 6 weeks post-partum and 1 year post partum
  Neonatal weight for height will be plotted from birth and at study visits up to 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Hoskin, R.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836